CLINICAL TRIAL: NCT03662997
Title: A Prospective, Randomized, Controlled Study Using Cross-Over Design to Evaluate and Compare 3 Multi-Layered Foam Dressings for the Management of Chronic Wounds
Brief Title: Clinical Study to Compare 3 Multi-Layered Foam Dressings for the Management of Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MxBFlex02
Record Dates: First submitted 2018-05-04; First posted 2018-09-10 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-01

CONDITIONS: Chronic Wound; Venous Leg Ulcer; Diabetic Foot Ulcer
Keywords: Chronic wound; Venous Leg Ulcer; Diabetic Foot Ulcer; Wound dressing
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: This is a prospective RCT using a crossover design to evaluate safety and efficacy. The study will be conducted in an outpatient setting of an academic clinical center. There will be two participant groups: those with VLU and those with DFU. Approximately 50% of the participants will be in the VLU group and 50% of the participants in the DFU group. Treatment sequence will be randomized so that a fair distribution is achieved. Each participant will receive a 2-week treatment with one of the three dressings followed by a 2-week treatment period with a second dressing (i.e. each participant will receive treatment with two different dressings, either the Bordered Five-Layer Foam Dressing and the Hydropolymer Foam Dressing, or the Bordered Five-Layer Foam Dressing and the Hydrocellular Multi-Layer Foam Dressing) using a cross-over (repeated measures) design, with a total of four study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Five-layer vs Hydropolymer (Active Comparator): Bordered Five-layer Foam Dressing for 2 weeks, followed by Hydropolymer Foam Dressing for 2 weeks.
  Interventions: Device: Bordered Five-Layer Foam Dressing; Device: Hydropolymer Foam Dressing
- Hydropolymer vs Five-layer (Active Comparator): Hydropolymer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  Interventions: Device: Bordered Five-Layer Foam Dressing; Device: Hydropolymer Foam Dressing
- Five-layer vs Hydrocellular (Active Comparator): Bordered Five-layer Foam Dressing for 2 weeks, followed by Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks.
  Interventions: Device: Bordered Five-Layer Foam Dressing; Device: Hydrocellular Multi-Layer Foam Dressing
- Hydrocellular vs Five-layer (Active Comparator): Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  Interventions: Device: Bordered Five-Layer Foam Dressing; Device: Hydrocellular Multi-Layer Foam Dressing

INTERVENTIONS:
Device: Bordered Five-Layer Foam Dressing — Bordered, five-layer, flexible foam dressing with soft silicone adhesive technology
  Other Names: Five-layer
Device: Hydropolymer Foam Dressing — Hydropolymer, adhesive foam island dressing
  Other Names: Hydropolymer
  Arms: Five-layer vs Hydropolymer; Hydropolymer vs Five-layer
Device: Hydrocellular Multi-Layer Foam Dressing — Multi-layered, hydrocellular foam dressing with silicone adhesive
  Other Names: Hydrocellular
  Arms: Five-layer vs Hydrocellular; Hydrocellular vs Five-layer

SUMMARY:
A prospective, randomized, controlled clinical trial (RCT) using a cross-over (repeated measures) design to evaluate safety and efficacy of three foam wound dressings in the local management of chronic wounds.

DETAILED DESCRIPTION:
The study will be conducted in an outpatient setting of an academic clinical center over a total period of four weeks (28 days, -1/+2).

The aim of this RCT is to evaluate and compare three different foam dressings in the local management of chronic wounds (i.e. venous leg ulcers (VLUs) and diabetic foot ulcers (DFUs)) in an outpatient setting. A bordered, five-layer, flexible foam dressing with soft silicone adhesive technology will be evaluated versus a hydropolymer, adhesive foam island dressing and a multi-layered, hydrocellular foam dressing with silicone adhesive, within three focus areas; efficacy and safety of the dressings, participant-centric outcomes and health economic evaluation.

Note: The terms used within the body of this report and results, in both the Primary and Secondary Outcomes, are defined as follows:

Period 1: Weeks 1 and 2 of study follow-up visits. Period 2: Weeks 3 and 4 of study follow-up visits. Week 1: Designates data captured only on visit days 7 and 21. Week 2: Designates data captured only on visit days 14 and 28. During Week 1: Designates data captured on visit days 3, 7, 17 and 21. During Week 2: Designates data captured on visit days 10, 14, 24 and 28. Day 3 of Week 1 from tables: inclusive of data captured on Visit Days 3 and 17. Day 3 of Week 2 from tables: inclusive of data captured on Visit Days 10 and 24.

Day 7 of Week 1 from tables: inclusive of data captured on Visit Days 7 and 21. Day 7 of Week 2 from tables: inclusive of data captured on Visit Days 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18-85 years of age with leg and foot ulcers (i.e. VLU, DFU).
2. Signed informed consent.
3. Subject and/or caregiver must be willing and able to tolerate multi-layered compression bandages when applicable and offloading footwear.
4. Study subject must be available and able to visit the clinic weekly for the full 4-week period.

Exclusion Criteria:

1. Pressure ulcers should not be included. Pressure injury as defined by the National Pressure Ulcer Advisory Panel (NPUAP).
2. Presence of local wound infection as determined by study doctor based on clinical signs and symptoms.
3. Subject has any evidence of peripheral arterial disease (PAD).
4. Subject diagnosed with malignancy other than cutaneous basal cell carcinoma.
5. Subject has received growth factor therapy (e.g. autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix e.g. amnion, amniotic tissue) within 2 weeks of screening date.
6. Pregnancy or lactation at time of study participation.
7. Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
8. Subject is currently enrolled or participated in another investigational device, drug or biological trial within 30 days of baseline of this study.
9. Present history of alcohol or drug abuse.
10. Known allergy/hypersensitivity to any of the components of the dressing.
11. Subject not suitable for the investigation according to the investigator's judgment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Alvarez, Principal Investigator — Vascular and Wound Care Center, University Hospital, Newark, NJ, USA
Locations (5):
- United States (5):
  - Center for Clinical Research, Inc., Castro Valley, California
  - Center for Clinical Trials, Inc., San Francisco, California
  - Vascular and Wound Care Center, Newark, New Jersey
  - SerenaGroup Research Foundation, Pittsburgh, Pennsylvania
  - SerenaGroup, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants were randomized and received treatment.
Groups:
- Hydropolymer vs Five-layer: Hydropolymer Foam Dressing for 2 weeks, then Bordered Five-Layer Foam Dressing for 2 weeks
- Five-layer vs Hydropolymer: Bordered Five-Layer Foam Dressing for 2 weeks, then Hydropolymer Foam Dressing for 2 weeks
- Hydrocellular vs Five-layer: Hydrocellular Multi-Layer Foam Dressing for 2 weeks then Bordered Five-Layer Foam Dressing for weeks
- Five-layer vs Hydrocellular: Bordered Five-Layer Foam Dressing for two weeks then Hydrocellular Multi-Layer Foam Dressing for two weeks
Period: Overall Study
Arm/Group | Hydropolymer vs Five-layer | Five-layer vs Hydropolymer | Hydrocellular vs Five-layer | Five-layer vs Hydrocellular
Started | 11 | 10 | 11 | 8
Completed | 11 | 8 | 11 | 8
Not Completed | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydropolymer vs Five-layer | Five-layer vs Hydropolymer | Hydrocellular vs Five-layer | Five-layer vs Hydrocellular | Total
Number analyzed (Participants) | 11 | 8 | 11 | 8 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 8 | 6 | 26
  >=65 years | 5 | 2 | 3 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 3 | 12
  Male | 8 | 6 | 7 | 5 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 11 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: % of Participants With Equal or Better Rate of Dressing Durability
Description: Dressing strike-through determined @ Wk1 Day 3&7, and Wk3 Day 17&21. Dressing strike-through that occurred Day 3 and/or 7, Day 17 and/or 21 were included in final dataset.
  Contributing factors to strike-through:
  Saturation of dressing pad:
  * Inappropriate dressing type
  * Inappropriate dressing change freq. (i.e. more frequent changes required)
  * Change in wound condition (e.g. increase in exudate amt)
  Dislodgement of dressing:
  * Suboptimal dressing application (e.g. selection of inappropriate dressing size, failure to clean periwound skin before applying dressing, insufficient fixation)
  * Exposure of dressing to mechanical forces (e.g. off-loading devices, patient mobility)
  * Patient interference w/ dressing
  Dressing design deficiency:
  * Insufficient fluid handling capacity (absorption, retention and/or moisture vapor transmission)
  * Insufficient adhesion
  * Insufficient conformability (i.e. ability to conform to body contours & challenging anatomical wound locations)
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting and analysis in order to compare # of incidences of strike-through when participants received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Groups:
- Five-layer vs Hydropolymer: The following two arms were combined into one cohort:
  1. Hydropolymer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Hydropolymer Foam Dressing for 2 weeks
- Five-layer vs Hydrocellular: The following two arms were combined into one cohort:
  1. Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Weeks 1 & 3 Five-layer equal or better | 100.0 | 94.1
  Weeks 2 & 4 Five-layer equal or better | 69.2 | 73.3
Statistical Analysis 1: Comparison: Five-layer vs Hydrocellular; Test type: Superiority — In this superiority study the primary efficacy analysis included constructing a two sided 5% significance level, using Fisher's non-parametric permutation test for ordered categorical variables and dichotomous variables for the differences. Numbers, percentages improved, not changed, worsened were analyzed with Mantel-Haenszel Exact Chi square over the course of 4 weeks in a 2x2 weeks treatment period inferiority will be established; p = 0.046, Chi-squared — Five-layer vs Hydrocellular arm, Weeks 1 & 3; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups
Statistical Analysis 2: Comparison: Five-layer vs Hydrocellular; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.56, Chi-squared — Five-layer vs Hydrocellular arm; Weeks 2 & 4; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups
Statistical Analysis 3: Comparison: Five-layer vs Hydropolymer; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.010, Chi-squared — Five-layer vs Hydropolymer arm; Weeks 1 & 3; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups
Statistical Analysis 4: Comparison: Five-layer vs Hydropolymer; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.25, Chi-squared — Five-layer vs Hydropolymer arm; Weeks 2 & 4; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups

2. Primary Outcome: % of Participants With No Strike-through After 7 Days Wear Time at Day 7 and 21
Description: Intact dressing after 7 days wear time, assessed @ Wk1 Day7 & Wk3 Day21 only. 1st week of dressing wear (Wks 1 & 3) is critical for start of wound healing.
  Contributing factors to strike-through:
  Saturation of dressing pad:
  * Inappropriate dressing type
  * Inappropriate dressing change freq. (i.e. more frequent changes required)
  * Change in wound condition (e.g. increase in exudate amt)
  Dislodgement of dressing:
  * Suboptimal dressing application (e.g. selection of inappropriate dressing size, failure to clean periwound skin before applying dressing, insufficient fixation)
  * Exposure of dressing to mechanical forces (e.g. off-loading devices, patient mobility)
  * Patient interference w/ dressing
  Dressing design deficiency:
  * Insufficient fluid handling capacity (absorption, retention and/or moisture vapor transmission)
  * Insufficient adhesion
  * Insufficient conformability (i.e. ability to conform to body contours & challenging anatomical wound locations)
Time Frame: Weeks 1 and 3
Population: as for outcome 1
Measure: Number; unit: %participants
Groups:
- Five-layer vs Hydropolymer: This arm was divided into 2 treatment groups:
  1. Hydropolymer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Hydropolymer Foam Dressing for 2 weeks
- Five-layer vs Hydrocellular: This arm was divided into 2 treatment groups:
  1. Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 14 | 18
%participants
  Five-layer | 43.8 | 35.3
  Comparator | 12.5 | 5.6
Statistical Analysis 1: Comparison: Five-layer vs Hydrocellular; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.046, Chi-squared, Corrected — Five-layer vs Hydrocellular; End of Weeks 1 and 3; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups
Statistical Analysis 2: Comparison: Five-layer vs Hydropolymer; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.010, Chi-squared, Corrected — Five-layer vs Hydropolymer; End of Weeks 1 & 3; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups

3. Secondary Outcome: % of Participants With Equal or Better Outcomes on Local Wound and Skin Pain Before Dressing Removal With Five-layer
Description: Pain was measured by subjects' responses to Visual Analogue Scale (VAS) of 0-10 at intervals of 2, 0=no pain, 10=worst pain ever.
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting and analysis in order to compare level of local wound and skin pain among participants who received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Five-layer equal or better | 92.3 | 75.1
  Week 2&4 Five-layer equal or better | 100.0 | 83.4

4. Secondary Outcome: % of Participants With Equal or Better Outcomes on Local Wound and Skin Pain at Removal With Five-layer
Description: as for outcome 3
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting & analysis in order to compare level of local wound and skin pain among participants who received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Fiver-layer equal or better | 69.3 | 87.6
  Week 2&4 Five-layer equal or better | 100.0 | 58.3

5. Secondary Outcome: % of Participants With Equal or Better Outcomes on Local Wound and Skin Pain Immediately After Dressing Removal With Five-layer
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Number; unit: %participants
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Five-layer equal or better | 77.0 | 81.3
  Week 2&4 Five-layer equal or better | 90.9 | 58.4

6. Secondary Outcome: % of Participants With Equal or Better Outcomes With Five-layer in Evaluation of the Dressings
Description: Dressing evaluation was determined via visual observation by study clinicians and categorized by saturation level: Partly saturated, Mostly saturated, and Strike-through.
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting & analysis in order to compare level of saturation in the dressings among participants who received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Five-layer equal or better | 100.0 | 70.6
  Week 2&4 Five-layer equal or better | 84.6 | 73.3

7. Secondary Outcome: % of Participants With Equal or Better Outcomes With Five-Layer When Assessing Wound Granulation
Description: Wound granulation was measured by visual assessment and photodigital planimetry. Wound granulation were grouped into 6 categories: None, <25%, 25-49%, 50-74%, 75-99%, 100%.
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting & analysis in order to compare level of wound granulation among participants who received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Groups:
- Five-layer vs Hydropolymer: This arm was divided into 2 treatment groups:
  1. Hydropolymer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Hydropolymer Foam Dressing for 2 weeks.
  Bordered Five-Layer Foam Dressing: Bordered, five-layer, flexible foam dressing with soft silicone adhesive technology
  Hydropolymer Foam Dressing: Hydropolymer, adhesive foam island dressing
- Five-layer vs Hydrocellular: This arm was divided into 2 treatment groups:
  1. Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
  2. Bordered Five-layer Foam Dressing for 2 weeks, followed by Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks.
  Bordered Five-Layer Foam Dressing: Bordered, five-layer, flexible foam dressing with soft silicone adhesive technology
  Hydrocellular Multi-Layer Foam Dressing: Multi-layered, hydrocellular foam dressing with silicone adhesive
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Five-layer equal or better | 92.3 | 93.8
  Week 2&4 Five-layer equal or better | 81.8 | 66.7

8. Secondary Outcome: % of Participants With Equal or Better Outcomes With Five-Layer When Assessing Wounds for Non-viable Tissue (Eschar, Fibrin Slough, Both)
Description: Non-viable tissue was determined by visual assessment and photodigital planimetry. Non-viable tissues were grouped into 5 categories: None, <25%, 25-49%, 50-74%, 75-100%.
Time Frame: 4 weeks
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting & analysis to compare the amount of non-viable tissue in the wound among participants who received one dressing or the other first for the 4 week treatment phase. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participants
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 16 | 18
%participants
  Week 1&3 Five-layer equal or better | 100.0 | 93.8
  Week 2&4 Five-layer equal or better | 90.9 | 91.6

9. Secondary Outcome: Mean Difference in Score in SF12 Health-Related Quality-of-Life Questionnaire
Description: The SF-12 health survey consists of 12 questions that yield an eight-scale profile of functional health and well-being, and 2 component summary measures of physical and mental health. SF-12 scores range from 0 to 100 with lower scores indicate lower levels of health.
  SF-12 questionnaire was administered at Screening/Baseline, Day 14, and Day 28 visits, and scored by a 3rd party vendor.
  Results are mean differences between five-layer vs the comparator dressing and presented for each of the 8 health domains, and 2 component summary measures.
  Negative scores indicate lower SF-12 scores (indicating lower levels of health) for the five-layer treatment group; positive scores indicate higher SF-12 scores for the five-layer group.
Time Frame: 4 weeks
Population: ITT analysis set. Means and standard deviations represent participants' responses from follow-up visits aggregated. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting & analysis in order to compare health-related quality-of-life when using each type of dressing. Number of participants analyzed differ from baseline due to missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 14 | 18
score on a scale
  Change in Physical Functioning | -0.896 (9.386) | -3.13 (13.84)
  Change in Role Physical | 1.99 (10.47) | 0.001 (11.461)
  Change in Bodily Pain | -6.57 (9.80) | 5.11 (14.31)
  Change in General Health | -0.449 (5.788) | 3.47 (9.89)
  Change in Physical Component | -0.545 (7.777) | 1.00 (10.06)
  Change in Role Emotional | -6.26 (12.68) | -2.61 (5.35)
  Change in Social Functioning | -7.12 (15.19) | -0.661 (18.685)
  Change in Vitality | -0.767 (14.391) | 2.63 (12.72)
  Change in Mental Health | -2.70 (7.70) | 0.395 (9.036)
  Change in Mental Component | -4.61 (9.35) | 0.078 (9.964)

10. Post Hoc Outcome: % Participant Compliance in Wear Time Between Five-layer and Comparator Dressing
Description: Compliance with the 7-day wear time protocol, within the first critical week of treatment.
  Compliance is defined as participants who wore a dressing continuously from time of application until removal at Day 7 visit. This includes participants whose dressing did not have strikethrough up to Day 7 and those who wore their dressing until strikethrough at Day 7 when dressing was removed.
Time Frame: 1 week
Population: Intent-to-treat (ITT) analysis set of superiority. Participants were combined into 2 cohorts: participants in the Five-layer vs Hydropolymer into one cohort, & Five-layer vs Hydrocellular were similarly combined into a second cohort to allow for reporting and analysis in order to compare the % of participant in compliance with 7-day wear time protocol in the first week of treatment. Number of participants analyzed differ from baseline due to missing values.
Measure: Number; unit: %participant
Arm/Group | Five-layer vs Hydropolymer | Five-layer vs Hydrocellular
Number analyzed (Participants) | 14 | 18
%participant
  First week compliance rate - Five-layer | 52.9 | 62.6
  First week compliance rate - Comparator | 27.8 | 18.8
Statistical Analysis 1: Comparison: Five-layer vs Hydrocellular; Test type: Superiority — This secondary outcome measure was not planned for at the initiation of the study. Compliance rates were calculated by combining the number incidences that dressings were worn for the full 7 days and when the dressings do not have strike-through during first the week of treatment; p < 0.05, Chi-squared — Five-layer vs Hydrocellular arm, first week of treatment; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups
Statistical Analysis 2: Comparison: Five-layer vs Hydropolymer; Test type: Superiority — This secondary outcome measure was not planned for at the initiation of the study. Compliance rates were calculated by combining the number incidences that dressings were worn for the full 7 days and when the dressings do not have strike-through during the first week of treatment; p < 0.05, Chi-squared — Five-layer vs Hydropolymer, first week of treatment; All data presented on the performance of the dressings reflect the FAS populations for the study comparison groups

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention.
Description: Safety population included all participants who received at least one dressing.
Groups:
- Hydropolymer, Then Five-layer: Hydropolymer Foam Dressing for 2 weeks, followed by Bordered Five-layer Foam Dressing for 2 weeks
- Five-layer, Then Hydropolymer: Bordered Five-layer Foam Dressing for 2 weeks, followed by Hydropolymer Foam Dressing for 2 weeks
- Hydrocellular, Then Five-layer: Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks followed by Bordered Five-layer Foam Dressing for 2 weeks
- Five-layer, Then Hydrocellular: Bordered Five-layer Foam Dressing for 2 weeks, followed by Foam Hydrocellular Multi-layer Foam Dressing for 2 weeks
Arm/Group | Hydropolymer, Then Five-layer | Five-layer, Then Hydropolymer | Hydrocellular, Then Five-layer | Five-layer, Then Hydrocellular
All-Cause Mortality (participants affected / at risk) | 1/11 | 4/9 | 0/11 | 1/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 4/9 | 0/11 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydropolymer, Then Five-layer (N=11) | Five-layer, Then Hydropolymer (N=9) | Hydrocellular, Then Five-layer (N=11) | Five-layer, Then Hydrocellular (N=9)
Blister plantar midfoot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain due to compression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased pain to study limb (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection to study ulcer (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blister left plantar forefoot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT03662997/Prot_SAP_000.pdf